CLINICAL TRIAL: NCT07076329
Title: Microbiota-Inflammation-Brain Axis in Heart Failure: New Food, biomarkerS and Artificial Intelligence Approach for the Prevention of undeRnutrition in Older
Brief Title: Microbiota-Inflammation-Brain Axis in Heart Failure: New Functional Food for the Prevention of undeRnutrition in Older
Acronym: AMBROSIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: University of Florence (Other); Northumbria University (Other); Synbiotec Srl (Industry); University College Dublin (Other); Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19882_spe
Record Dates: First submitted 2025-06-17; First posted 2025-07-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation (AF); Heart Failure
Keywords: gut microbiota; elderly; probiotics; functional food; frailty; inflammation; heart failure; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Frailty; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambrosia group (Experimental): Participants in the intervention group will receive the AMBROSIA Bar along with standard nutritional counselling. The AMBROSIA Bar is a functional chocolate-based food product designed specifically for older adults with heart failure and/or atrial fibrillation. It contains a tailored blend of ingredients, including:
  Probiotic strains (Lacticaseibacillus rhamnosus Istituto Microbiologico C. N. R.501® and Lacticaseibacillus paracasei Istituto Microbiologico C. N. R.502®, branded as SYNBIO®), Hydrolysed proteins, Inulin (a dietary fiber), Coenzyme Q10
  Participants will consume one AMBROSIA Bar per day for 6 months. The formulation aims to support muscle health, improve nutrient absorption, modulate the gut microbiota, and reduce inflammation.
  Interventions: Dietary Supplement: Ambrosia bar
- Control group (No Intervention): Participants in the control group will receive standard nutritional counseling.

INTERVENTIONS:
Dietary Supplement: Ambrosia bar — The experimental intervention involves the "AMBROSIA" bar alongside healthy dietary counseling.
  The "AMBROSIA" bar is a novel chocolate bar designed for older Heart Failure (HF) and Atrial Fibrillation (AF) patients to prevent undernutrition. Its distinguishing features are:
  * Unique Composition: It contains a unique and specific blend of probiotic strains and a cocktail of micro/macronutrients.
  * Patented Probiotic Efficacy: The SYNBIO® blend is patented (RM2004A000166, EP1743042) for its exceptional intestinal mucosal adhesion, ensuring effective colonization and persistence.
  * Optimal Delivery Matrix: The chocolate bar serves as a palatable and effective vehicle for probiotic delivery, confirmed to maintain probiotic viability.
  * Targeted Nutritional Strategy: The bar aims to modulate gut microbiota and address undernutrition, inflammation, and cachexia in the target.
  Arms: Ambrosia group

SUMMARY:
The goal of this clinical trial is to learn if the AMBROSIA Bar helps prevent undernutrition and muscle loss in older adults with heart failure or atrial fibrillation.

The main questions it aims to answer are:

Does the AMBROSIA Bar help improve muscle mass and physical performance in older adults with heart conditions? What effects does the AMBROSIA Bar have on body composition, quality of life, inflammation, nutrition status, and gut microbiota?

Researchers will compare people who assume the AMBROSIA Bar in addition to nutritional counseling to those who only receive nutritional counseling.

Participants will:

* Receive nutritional counseling and consume one AMBROSIA Bar per day for 6 months (intervention group) or receive nutritional counseling only (control group).
* Receive clinical assessment at the moment of enrolment, after 3 months, and after 6 months
* Give samples (blood, saliva, urine, and stool) and complete questionnaires to check their nutrition, cognitive, and physical health

ELIGIBILITY:
Inclusion Criteria:

* Age >70 years;
* Caucasian ethnicity;
* Diagnosis of atrial fibrillation (AF) and/or heart failure (HF);
* Normal nutritional status or at risk of malnutrition;
* Adherence to Mediterranean diet

Exclusion Criteria:

* Obesity (BMI >30 Kg/m2);
* Underweight (BMI <18.5 Kg/m2);
* Use of antibiotics, corticosteroids and immune-suppressors in the last 6 months;
* Immunodeficiency;
* Trip to exotic areas in the last 12 months;
* Recent (<3 months) major surgical procedure;
* Uncontrolled diabetes mellitus;
* Active cancer;
* Chronic significant hepatic diseases;
* Chronic renal failure (KDIGO stages 4-5);
* Dementia and severe mental diseases;
* Other conditions interfering with autonomous drugs assumption;
* Chronic use of NSAIDs;
* Relevant history of allergy or infectious diseases

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Skeletal Muscle Mass at 6 months | From enrollment to the end of treatment at 6 months.
  A change in skeletal muscle mass from baseline versus the control group as assessed by Bioelectrical Impedence Analysis, change in physical performance as evaluated with SHORT PHYSICAL PERFORMANCE BATTERY test, a measure of frailty).

SECONDARY OUTCOMES:
Changes to anthropometry | From enrollment to the end of treatment at 6 months.
  Weight (kg) and height (m) will be measured and used to calculate Body Mass Index (BMI, kg/m²). Each parameter will be analyzed separately.
Changes to body composition | From enrollment to the end of treatment at 6 months.
  Change in body composition assessed by Bioelectrical Impedance Analysis (BIA): Fat Mass (FM, kg), Fat Free Mass (FFM, kg), and Body Cell Mass (BCM, kg). In addition, FFM will be combined with height (m) to calculate Fat-Free Mass Index (FFMI, kg/m²). Each parameter will be reported and analyzed separately.
Impacts on Quality of Life associated with Bowel Function: | From enrollment to the end of treatment at 6 months.
  Changes in quality of life assessed by Gastrointestinal Quality of Life Index (GIQLI). The GIQLI is a validated 36-item questionnaire measuring gastrointestinal-specific quality of life. Scores range from 0 to 144. Higher scores indicate better quality of life..
Change in Geriatric Depression Scale (GDS-15) score | From enrollment to the end of treatment at 6 months.
  The GDS-15 is a self-report screening tool for depression in older adults. Scores range from 0 to 15; higher scores indicate more severe depressive symptoms.
Change in Mini-Mental State Examination (MMSE) score | From enrollment to the end of treatment at 6 months.
  The MMSE is a cognitive screening tool scored from 0 to 30. Higher scores indicate better cognitive function.
Change in handgrip strength | From enrollment to the end of treatment at 6 months.
  Measured using a hand dynamometer. Results expressed in kilograms (kg). Higher values indicate better muscle strength.
Change in Clinical Frailty Scale (CFS) | From enrollment to the end of treatment at 6 months.
  Assessed using the Clinical Frailty Scale, a 9-point scale (1 = very fit; 9 = terminally ill). Higher scores indicate worse frailty.
Impacts on the composition of the fecal microbiota | From enrollment to the end of treatment at 6 months.
  Evaluation of changes in the gut microbiota profile through 16s RNA targeted sequencing.
Changes to nutritional and inflammatory biomarkers in blood samples | From enrollment to the end of treatment at 6 months.
  Changes in circulating inflammatory markers, mainly plasma cytokine profiles, and blood markers of undernutrition, using the immunoassays based on Luminex xMAP (multi-analyte profiling) technology which enable simultaneous detection and quantification of multiple secreted proteins.
Changes to blood lipid profile | From enrollment to the end of treatment at 6 months.
  Modifications in the blood lipid profile, using gas chromatography techniques.
Modifications in metabolomic profiles in plasma, saliva, and stool samples. | From enrollment to the end of treatment at 6 months.
  Metabolite profiles of plasma, urine and faecal water in all samples will be generated through reverse phase (plasma) and hydrophilic interaction (urine, faecal water) chromatography, in order to define potential markers of undernutrition and responsiveness to nutritional intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT07076329/Prot_ICF_000.pdf